CLINICAL TRIAL: NCT01280396
Title: Metabolic Side-effects in Patients Receiving Clozapine and Second-generation Antipsychotics in an Outpatient Clinic
Brief Title: Metabolic Side-effects for Second-generation Antipsychotics
Status: Completed | Type: Observational
Sponsor: The University of Hong Kong (Other)
Collaborators: Queen Mary Hospital, Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Albert Kar-Kin Chung, Clinical Assistant Professor, The University of Hong Kong
Other Study IDs: HKCTR-1205
Record Dates: First submitted 2011-01-19; First posted 2011-01-20 (Estimated); Last update posted 2018-05-03 (Actual); Status verified 2018-04

CONDITIONS: Mental Disorders
Keywords: metabolic; SGAs; clozapine
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- SGAs: patients receiving SGAs

SUMMARY:
Second-generation antipsychotics (SGAs), including clozapine, are commonly used nowadays as treatment for psychosis. There are increasing concerns about their related metabolic side-effects over weight gain, risks to cause glucose intolerance and hyperlipidemia, and a specific condition known as metabolic syndrome. All these side-effects might be associated with the increased risk of cardiovascular diseases and diabetes mellitus.

This study is to analyze the simple physical measurements (weight and height) and venous blood tests (for fasting blood glucose and lipid) results collected routinely since 2008 (recommended by the local hospital authority as a territory-wide "SGAs Monitoring Program") from those outpatients receiving SGAs (amisulpride, aripiprazole, olanzapine, paliperidone, quetiapine, risperidone and ziprasidone) and/or clozapine, at a local psychiatric outpatient clinic in Hong Kong. The investigators hypothesized that there should be differential risks on metabolic side-effects amongst these SGAs.

ELIGIBILITY:
Inclusion Criteria:

* was ≥18 years of age
* out-patients
* had received any one of these antipsychotics: aripiprazole, amisulpride, clozapine, olanzapine, paliperidone, quetiapine, risperidone, ziprasidone
* consented to provide physical measurements and venous blood samples

Exclusion Criteria:

* not consented to provide venous blood samples and/or physical measurement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Out-patients in a public psychiatric out-patient centre
Sampling Method: Non-Probability Sample
Enrollment: 241 (Actual)
Dates: Start 2010-11; Primary Completion 2012-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
development of metabolic syndrome according to IDF criteria | 1 year
  post treatment with second generation antipsychotics

SECONDARY OUTCOMES:
change in BMI | 1 year
  post treatment with second generation antipsychotics

CONTACTS AND LOCATIONS:
Overall Officials: Albert Kar Kin Chung, MBBS, Principal Investigator — Department of Psychiatry, Queen Mary Hospital
Locations (1):
- Western Psychiatric Centre, Hong Kong, Hong Kong